CLINICAL TRIAL: NCT02123342
Title: Promoting Exercise Among Older Malaysians Using SMS Reminders. The Malaysian Physical Activity for Health Study (myPAtHS): A Randomized Controlled Trial
Brief Title: SMS Reminders for Exercise Among Older Adults. Malaysian Physical Activity for Health Study
Acronym: myPAtHS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UM.C/625/1/HIR/MOHE/ASH/02-PA
Record Dates: First submitted 2014-04-20; First posted 2014-04-25 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Physical Activity; Exercise
Keywords: health; older adults; mobile phone
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Exercise programme only (No Intervention): Participants randomized in this condition will not receive SMS reminders to execute the myPAtHS exercise programme.
- SMS reminder (Experimental): Participants in this study arm will receive SMS reminders to motivate them to execute the myPAtHS exercise programme.
  Interventions: Behavioral: Exercise programme plus SMS reminders

INTERVENTIONS:
Behavioral: Exercise programme plus SMS reminders — Participants will receive SMS reminders for their myPAtHS exercise programme compared to the other group where participants will only receive the myPAtHS exercise programme.
  Arms: SMS reminder

SUMMARY:
The purpose of the study is:

1) To evaluate the efficacy and feasibility of an SMS reminder intervention for promoting an health-related exercise programme (myPAtHS) among older Malaysian adults, in a randomized controlled trial (RCT).

Hypothesis: Frequency and duration of the exercise programme execution will be higher for the SMS reminder condition compared to the programme only condition. The effect may be reduced from post- to follow-up measurement (24 weeks after baseline and 12 weeks after post-measurement) but all outcomes will remain significantly higher at 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Mobile phone user
* Acceptable health that does not prevent exercise
* Acceptable command of the English language
* No engagement in a regular- structured exercise routine like gym training or other structured programmes
* Interest in an exercise programme
* Willing to attend scheduled follow-up sessions at 12 weeks (pre-post evaluation) and 24 weeks (post-intervention evaluation) after the first session

Exclusion Criteria:

* participants who have any medical condition or health concern that would restrict regular exercise based on one screening question. If this question will be answered with "yes" participants are advised to seek medical care.

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Number of myPAtHS exercise sessions. | 12 weeks & 24 weeks
  This will be assessed with an exercise diary.
Time spent doing the myPAtHS exercise programme. | 12 weeks & 24 weeks
  This will be assessed with an exercise diary.

SECONDARY OUTCOMES:
Change in overall physical activity. | baseline, 12 weeks & 24 weeks
  The International Physical Activity Questionnaire (short version) will be used to collect physical activity data.
Change in exercise self-efficacy. | baseline, 12 weeks & 24 weeks
  The Exercise Self-Efficacy-Scale will be used to collect exercise self-efficacy data.
Change in grip strength. | baseline, 12 weeks & 24 weeks
  Grip strength will be assessed using the North Coast strength dynamometer (North Coast Hydraulic Hand Dynamometer, North Coast Medical Inc, Morgan Hill, California, USA).
Change in leg-strength. | baseline, 12 weeks & 24 weeks
  Leg-strength will be collected using the 30 seconds chair-stand-test.
Subjective intensity while doing the myPAtHS exercise programme. | 12 weeks & 24 weeks
  This will be assessed with an exercise diary.

CONTACTS AND LOCATIONS:
Overall Officials: ANDRE M MüLLER, MA, Principal Investigator — University of Malaya; SELINA KHOO, PhD, Study Chair — University of Malaya; TONY MORRIS, PhD, Study Chair — Victoria University
Locations (1):
- Premises of research participants, Petaling Jaya, Selangor, Malaysia

REFERENCES:
- [Derived] Muller AM, Khoo S, Morris T. Text Messaging for Exercise Promotion in Older Adults From an Upper-Middle-Income Country: Randomized Controlled Trial. J Med Internet Res. 2016 Jan 7;18(1):e5. doi: 10.2196/jmir.5235. PMID 26742999